CLINICAL TRIAL: NCT01355939
Title: A Prospective Multicenter Trial to Evaluate Adhesion Characteristics and Adhesiolysis-related Complications of Barrier-coated and Non-barrier-coated Intraperitoneal Mesh During Abdominal Re-exploration After Prior Ventral Hernia Repair
Brief Title: Comparative Effectiveness Multicenter Trial for Adhesion Characteristics of Ventral Hernia Repair Mesh
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-02112; 1KM1CA156708-01 (NIH)
Record Dates: First submitted 2011-04-26; First posted 2011-05-19 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Ventral Hernia; Adhesions
Keywords: Hernia; Adhesiolysis; Adhesions; Intraperitoneal Mesh; Abdominal Re-exploration; Mesh; Barrier-Coated Mesh; Non-Barrier-Coated Mesh; Laparoscopic Approach; Open Approach; Abdominal Re-Exploration Surgery
MeSH Terms: conditions — Hernia, Ventral; Tissue Adhesions; Hernia | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Abdominal surgery after prior VHR with barrier-coated mesh
  Interventions: Procedure: Clinically-Indicated Abdominal Re-Exploration Surgery
- Abdominal surgery after prior VHR with nonbarrier-coated mesh
  Interventions: Procedure: Clinically-Indicated Abdominal Re-Exploration Surgery
- Lap adhesiolysis during abdominal surgery after prior VHR
  Interventions: Procedure: Clinically-Indicated Abdominal Re-Exploration Surgery
- Open adhesioloysis during abdominal surgery after prior VHR
  Interventions: Procedure: Clinically-Indicated Abdominal Re-Exploration Surgery

INTERVENTIONS:
Procedure: Clinically-Indicated Abdominal Re-Exploration Surgery — This is a prospective observational study. Abdominal re-exploration surgery is clinically-indicated and planned as the standard of care for the patients regardless of their decision to participate in the study.
  Other Names: Bard(TM) Mesh; PROLENE(TM); ProLite(TM); ProLite(TM) Ultra(TM); Bard(TM) Soft Mesh; PROLENE(TM) Soft; Parietex(TM) Flat Sheet TEC; INFINIT(TM) Mesh; C-QUR Lite(TM); ULTRAPRO(TM); PROLENE(TM) Hernia System; Bard(TM) Mesh PerFix Plug; Bard(TM) Ventralex; C-QUR(TM) Mesh; PROCEED(TM); Bard(TM) Sepramesh(TM) IP Composite; Parietex(TM) Composite; PHYSIOMESH(TM); Bard(TM) Composix(TM) E/X; Bard(TM) Composix(TM) L/P; DUALMESH(R); DUALMESH(R) Plus; VICRYL(TM); TIGR(R) Matrix; Gore (R) Bio-A(R); AlloDerm(R); AlloMax(TM); FlexHD(R); Biodesign(TM) Surgisis(R); Strattice(TM); XenMatrix(TM); Veritas(R); SurgiMend(R); Peri-Guard(R); Permacol(TM); CollaMend(TM) FM; CollaMend(TM)

SUMMARY:
The proposed study will compare the benefits, harms, and comparative effectiveness of intraperitoneal barrier-coated and non-barrier coated ventral hernia repair (VHR) mesh in reducing adhesions, adhesion-related complications, and adhesiolysis sequelae in actual patient subpopulations and clinical circumstances. A subset of the data will be analyzed to compare the benefits, harms, and comparative effectiveness of the laparoscopic and open approaches to adhesiolysis. A comprehensive array of health-related risk factors and patient-centered outcomes will be assessed in the investigators diverse patient population for proper multivariate data analysis.

Specific Aim I: To evaluate and compare the adhesion characteristics of intraperitoneal barrier-coated versus non-barrier-coated mesh during abdominal re-exploration after prior ventral hernia repair.

Specific Aim II: To evaluate and compare the adhesion-related complications and adhesiolysis-related complications of intraperitoneal barrier-coated versus non-barrier-coated mesh during abdominal re-exploration after prior ventral hernia repair.

Specific Aim III: To determine the comparative effectiveness of intraperitoneal barrier-coated versus non-barrier-coated ventral hernia repair mesh in reducing adhesions, adhesion-related complications, and adhesiolysis sequelae in actual patient subpopulations and clinical circumstances.

Specific Aim IV: To evaluate and compare the adhesiolysis-related complications of the laparoscopic and open approaches to adhesiolysis during abdominal re-exploration after prior ventral hernia repair.

Specific Aim V: To determine the comparative effectiveness of the laparoscopic and open approaches to adhesiolysis during abdominal re-exploration after prior ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* prior ventral hernia repair with intraperitoneal placement of mesh (open or laparoscopic approach; absorbable barrier-coated mesh, permanent barrier-coated composite mesh, permanent barrier-coated noncomposite mesh, non-barrier-coated polypropylene mesh, or biologic mesh)
* subsequent abdominal procedure requiring exposure of entire surface area of intraperitoneal mesh

Exclusion Criteria:

* less than 18 years of age
* inability to verify intraperitoneal mesh type or location
* active abdominal wound infection or open abdominal wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators' patient population
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mesh adhesiolysis time:Mesh surface area | Intraoperatively (day 1)

SECONDARY OUTCOMES:
Mesh Contracture | Intraoperatively (day 1)
Mesh adhesion tenacity | Intraoperatively (day 1)
Percentage mesh surface area covered with adhesions | Intraoperatively (day 1)
Adhesiolysis time to abdominal wall | Intraoperatively (day 1)
Adhesiolysis time to mesh | Intraoperatively (day 1)
Incidence of adhesiolysis-related intra-operative complications | Intraoperatively (day 1)
Length of stay of hospital admission | 30 day postoperative
Length of stay in ICU | 30 day postoperative
Interval to return to bowel function | 30 day postoperative
Interval to return to independent ambulation or activities of daily living | 30 day postoperative
Interval to return to work or routine physical activity | 30 day postoperative
Incidence of postoperative complications | 30 day, 12 month, and 24 month postoperative
Incidence of surgical site infection | 30 day, 12 month, and 24 month postoperative
Incidence of initiation of antibiotics, blood and total parenteral nutrition | 30 day, 12 month, and 24 month postoperative
Incidence of bedside procedures to address a postoperative surgical complication | 30 day, 12 month, and 24 month postoperative
Incidence of surgery under local anesthesia to address a postoperative complication | 30 day, 12 month, and 24 month postoperative
Incidence of single system organ failure | 30 day, 12 month, and 24 month postoperative
Incidence of multiple-system organ failure | 30 day, 12 month, and 24 month postoperative
Mortality rate | 30 day, 12 month, and 24 month postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brunt, M.D., Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - University of California-San Diego, San Diego, California
  - Baystate Medical Center, Springfield, Massachusetts
  - Washington University, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Greenville Medical Center, Greenville, South Carolina